CLINICAL TRIAL: NCT06046612
Title: The Effect of Empagliflozin on Peripheral Microvascular Dysfunction in Heart Failure With
Brief Title: Empagliflozin for Peripheral Microvascular Dysfunction in Heart Failure With Preserved Ejection Fraction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20225016824500
Record Dates: First submitted 2023-04-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Microvascular Dysfunction
Keywords: Heart failure; Empagliflozin; Jardiance; microvascular disease; microvascular function
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Participants receive 10mg Empaglifozin once daily on prescription from their treating physician. This is not an intervention in this trial, but part of their normal HFpEF treatment.
  At the start of the study patients will undergo the LASCA measurements. A very small amount of acetylcholine, nitroprusside and insulin will be applied to the skin of the forearm, to stimulate the bloodflow during LASCA. After 3 months of use of Empagliflozin the LASCA measurement will be repeated. Furthermore, at each visit 4 tubes of blood will be drawn for biobanking, and patients will be asked to fill out a quality of life questionnaire. During the trial, patients will be monitored in routine clinical care as indicated by their treating physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- heart failure with preserved ejection fraction (Experimental): Empagliflozin 10mg, tablet, once daily
  Interventions: Drug: Participants receive 10mg Empaglifozin once daily on prescription from their treating physician. This is not an intervention in this trial, but part of their normal HFpEF treatment

INTERVENTIONS:
Drug: Participants receive 10mg Empaglifozin once daily on prescription from their treating physician. This is not an intervention in this trial, but part of their normal HFpEF treatment — The investigational medicinal product investigated in this trial (empagliflozin) is authorised for use in the European Union by the European Medicines Agency and will be used in accordance with the terms of the marketing authorization. The treating physician (cardiologist) will determine the indication for empagliflozin use, discuss the benefits and risks with the patient, prescribe the drug, and provide follow up after starting the drug, according to normal clinical practice. The study participants are not assigned to a particular therapeutic strategy decided by the clinical trial protocol.
  Other Names: Jardiance

SUMMARY:
The goal of this low-intervention clinical trial is to learn about the effect of the drug Empagliflozin in patients with heart failure with preserved ejection fraction.

The main questions it aims to answer are:

* What is the effect of treatment with Empagliflozin after 3 months on peripheral microvascular function
* Do clinical correlates for worse microvascular function exist, and thus identify patients that could possibly benefit most from empagliflozin treatment

Patients will use Empagliflozin, prescribed by their treating physician. Before the start of treatment and after 3 months they will be asked to

* Fill out a quality of life questionnaire
* Draw 4 tubes of blood
* Undergo non-invasive measurement of the blood flow of the microvasculature in the forearm (using laser speckle contrast analysis)

DETAILED DESCRIPTION:
Heart failure (HF) with preserved ejection fraction (HFpEF), is an important public health problem with a poor prognosis and many people are affected by it. Microvascular dysfunction (MVD) is thought to play an important role in this complex syndrome. MVD may lead to disease progression in HFpEF. For the past years the main focus of HFpEF treatment has been on symptom relieve and diagnosing and treating co-occurring disease, such as hypertension or diabetes. Recently, the sodium-glucose co-transporter 2 (SGLT-2) inhibitor Empagliflozin was suggested to be added to this list of treatments. This drug was proven to reduce the combined risk of cardiovascular death or HF hospitalization in HFpEF patients in the EMPEROR-PRESERVED trial. Preclinical studies have proposed an important role for microvascular function in the mechanism of action of empagliflozin in HFpEF. The microvasculature may also play an important role in the etiology of HFpEF.

The microcirculation in the skin is accessible and suitable for analysis of microvascular function. Laser speckle contrast analysis (LASCA) is a relatively new and non-invasive analysis that measures the blood flow in the skin microvasculature using several stimuli.

In HFpEF patients no clinical research has been conducted to evaluate the effect of Empagliflozin on MVD, despite its seemingly important role in the HFpEF etiology. We hypothesize that empagliflozin improves microvascular function in HFpEF patients. Understanding of the effects of this important drug in the treatment of HFpEF is essential to optimize its use in this growing population. Key clinical determinants may exist that improve our ability to determine which patients at what disease stage can specifically benefit from this intervention. The patients with the strongest improvement in MVD during treatment with Empagliflozin might benefit most regarding cardiac function or wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* HFpEF diagnosis according to the ESC 2021 Guidelines for the diagnosis and treatment of acute and chronic heart failure Symptoms and signs of HF LVEF ≥ 50% (on any imaging modality) Objective evidence of cardiac structural and/or functional abnormalities consistent with the presence of LV diastolic dysfunction/ raised LV filling pressures, including raised natriuretic peptides (table 1) OR invasively measured pulmonary capillary wedge pressure (PCWP) of >15 mmHg (at rest) or ≥25 mmHg (with exercise) or left ventricular end diastolic pressure ≥ 16 mmhg (at rest).
* Ability to understand and speak the Dutch language
* Treatment with empagliflozin 10mg once daily is planned to be started by the treating physician
* Signed informed consent

Exclusion Criteria:

* Unable or unwilling to sign informed consent
* Under 18 years of age
* Contra-indication to the use of empagliflozin Severe kidney disease (Glomerular filtration rate< 20 ml/min) Severe liver insufficiency Recent (<12 months) or planned major surgery (Including coronary artery bypass grafting, cardiac valve replacement) Severe acute disease (< 12 months) (Including acute coronary syndrome, TIA/CVA) Pregnancy
* Use of empagliflozin or other SGLT-2 inhibitor at baseline
* Known hypersensitivity to empagliflozin, acetylcholine, sodium nitroprusside or insulin
* Insulin dependent patients (Fasting conditions cause a risk of ketoacidosis in these patients).
* Subjects currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study.
* Any condition that interferes with the correct execution of the LASCA measurements (patient is unable to keep arms motionless during the measurements, any condition that does not allow disposables to be attached to the forearm skin)
* Any other reason that makes it undesirable for patient to use empagliflozin according to the researcher / treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-08-13 (Estimated); Study Completion 2025-02-13 (Estimated)

PRIMARY OUTCOMES:
Cutaneous vascular conductance (CVC) | Change from baseline to 3 months
  Skin blood flow (arbitrary perfusion units, APU) is divided by the mean arterial pressure to yield the CVC.

SECONDARY OUTCOMES:
baseline bloodflow and area under the curve | Change from baseline to after 3 months
  as measured by LASCA
Serum ketone levels in mmol/L | Change from baseline to after 3 months
  Serum ketone levels in mmol/L
EQ5D-5L questionnaire score | Change from baseline to 3 months
  index value, ranging from 1 to -0.5. a higher value is a better outcome analogue scale and single index value
EQ5D-5L questionnaire score | Change from baseline to 3 months
  visual analogue scale, ranging from 1 to 100, a higher value is a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Hospital, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mourmans SGJ, Achten A, Hermans R, Scheepers MJE, D'Alessandro E, Swennen G, Woudstra J, Appelman Y, Goor HV, Schalkwijk C, Knackstedt C, Weerts J, Eringa EC, van Empel VPM. The effect of empagliflozin on peripheral microvascular dysfunction in patients with heart failure with preserved ejection fraction. Cardiovasc Diabetol. 2025 Apr 25;24(1):182. doi: 10.1186/s12933-025-02679-8. PMID 40281528